CLINICAL TRIAL: NCT01002885
Title: The Use of FSH Receptor Polymorphisms To Improve Pregnancy Rates In In-Vitro Fertilization
Brief Title: Follicle Stimulating Hormone (FSH) Receptor Polymorphisms in In-Vitro Fertilization Cycles.
Status: Completed | Type: Observational
Sponsor: University Reproductive Associates (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Peter McGovern, MD, Director, University Reproductive Associates
Other Study IDs: 0120090163
Record Dates: First submitted 2009-10-26; First posted 2009-10-28 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Infertility
Keywords: Infertility; FSH Receptor Polymorphisms
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 EDTA containing lavender topped tubes will be collected before, during or within 3 months after an IVF cycle. Genomic DNA will be extracted and saved for genotyping.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is being done to identify if certain sequences (patterns) of key genes (called polymorphisms) may predict a response to fertility medications. The investigators will also determine if the individual response to fertility medications affects pregnancy rates in in-vitro fertilization.

DETAILED DESCRIPTION:
All IVF patients who meet inclusion criteria and not exclusion criteria will be asked to participate in this study. Upon consent, a blood sample will be obtained in 2 EDTA containing lavender topped tubes before, during or within 3 months after their IVF cycle. Genomic DNA will be extracted and saved for genotyping.

The Investigators will collect data on each individual's age, ethnic background, and estradiol levels on the day of hCG administration, total gonadotropin amount, clinical pregnancy rates, basal FSH levels, and occurrence of OHSS. The Investigators will then analyze all samples from all patients for their FSH receptor genotypes.

Patients will be compensated $75 via a check within 6-8 weeks of their blood drawn.

ELIGIBILITY:
Inclusion Criteria:

1. 100 women less than 35 years old at time of signing the Informed Consent Form.
2. Day 3 FSH level less than or equal to 10 mIU/ml with an estradiol < 70 pg/ml
3. Day 3 antral follicle count of greater than 10 follicles total.
4. Couples who have male factor infertility, tubal factor infertility, and unexplained infertility.

Exclusion Criteria patients who have:

1. Endometriosis
2. Polycystic ovarian syndrome

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing in-vitro fertilization will be recruited. Inclusion criteria will limit the patient population to those patients most likely to have normal ovarian function since age or disease related ovarian dysfunction will confound interpretation of our results.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2009-07; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is to evaluate the frequency of FSH receptor polymorphisms in our population. | 3 years
  The investigators are looking to quantify how often certain FSH receptor Polymorphisms occur in the population and cetain racial groups. We will be looking at patient's race along with the laboratory results.

SECONDARY OUTCOMES:
The secondary outcome is to further clarify the variation in response to FSH due to FSH receptor polymorphisms using the protocols largely used in the United States, including our center. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Seungdamrong, MD, Principal Investigator — University Reproductive Associates
Locations (2):
- United States (2):
  - University Reproductive Associates, Hasbrouck Heights, New Jersey
  - University Reproductive Associates, Hoboken, New Jersey